CLINICAL TRIAL: NCT03469102
Title: Diagnostic Value of 18FDG PET/CT Textural Indices in Patients With an Adrenal Lesion
Brief Title: 18FDG PET Textural Indices in Adrenal Lesion
Acronym: ImpactTexture
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: Impact Texture Surrénale
Record Dates: First submitted 2018-03-05; First posted 2018-03-19 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-03

CONDITIONS: Adrenal Tumor
Keywords: Positron emission tomography; Texture indices; Diagnostic performance
MeSH Terms: conditions — Adrenal Gland Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Tumors are characterized by a great heterogeneity. Characterizing this intra-tumor heterogeneity is a major challenge in oncology to improve the therapeutic management and move towards personalized medicine adapted to each patient. However, intra-tumor heterogeneity remains rarely used for diagnostic purposes The discovery of an adrenal mass can occur in different circumstances. Detection of an adrenal mass can be done in a context of secreting syndrome, in the assessment of an extra-adrenal neoplasia or fortuitously when performing an imaging for another reason. The etiologies are numerous (cortical tumors, medullary tumors, metastatic lesion of a extra-adrenal neoplasia, others). The adrenal masses can be divided into two categories, depending on whether they are hyperfunctional or not. In patients without an oncological history, an adrenal mass discovered is most often a benign adenoma, but requires an endocrine assessment. In patients with known primary cancer, approximately 30% of the adrenal masses are malignant.

In all cases, the diagnostic procedure includes an imaging assessment to characterize the lesion and an endocrine assessment. CT scan performed without and after intravenous iodinated contrast agent injection is the first-line examination to assess an adrenal mass.

18F-FDG-PET may be indicated as second-line for characterizing an adrenal mass. Adrenal tumor SUVmax (Standard Uptake Value) and adrenal tumor SUVmax / liver SUVmax ratio are routinely used to determine the malignancy of a lesion. Although very useful for assessing the glucose metabolism of a given lesion, these parameters do not allow assessing the heterogeneity of tumor uptake. The texture analysis corresponds to an analysis of the spatial distribution of FDG uptake, and allows, by the calculation of many indices, an evaluation of the heterogeneity of the tumors.

The hypothesis of our study is that the texture parameters could have an additional diagnostic value to improve the performance of conventional quantitative parameters to determine the malignancy of a lesion.

The objective of this study is to investigate the diagnostic value of texture indices in a large cohort of patients presenting an adrenal lesion

ELIGIBILITY:
Inclusion Criteria:

* Having benefited from a 18-FDG PET-CT scan in the nuclear medicine department of University Hospital of Brest
* Addressed in the context of an assessment of an adrenal lesion, in the evaluation of an extra-adrenal neoplasia or other motive
* presenting an adrenal lesion
* From June 29, 2012 to June 30, 2017

Exclusion Criteria:

* Patients followed in another center than the University Hospital of Brest
* Lesions of undetermined nature
* Diagnosis of benignity or malignancy not confirmed by anatomopathology.
* Patient having expressed his opposition to the use of his medical data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: presenting an adrenal lesion
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-27 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of FDG PET/CT textural indices | 6 months
  Area Under the Curve

SECONDARY OUTCOMES:
Cut off value of FDG PET/CT textural indices | 6 months
  For each cut off value : Sensibility(%)
Cut off value of FDG PET/CT textural indices | 6 months
  For each cut off value : Specificity(%)
Cut off value of FDG PET/CT textural indices | 6 months
  For each cut off value : Positive and Negative Predictive Value (%),
Cut off value of FDG PET/CT textural indices | 6 months
  For each cut off value : Accuracy (%)

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France